CLINICAL TRIAL: NCT01169597
Title: Short Term Study on the Effect of a Fixed Dose of 12.5 mg of Prednisone as Starting Dose in Polymyalgia Rheumatica
Brief Title: Short Term Efficacy of a Starting Dose of 12.5 mg of Prednisone in Polymyalgia Rheumatica Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Genova (Other)
Responsible Party: Prof. Marco A Cimmino, Dept. of Internal Medicine, University of Genova, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMR-PDN001
Record Dates: First submitted 2010-07-21; First posted 2010-07-26 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-06

CONDITIONS: Polymyalgia Rheumatica
Keywords: polymyalgia rheumatica; prednisone; clinical examination; remission; ultrasonography
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: prednisone — prednisone 12.5 mg daily po

SUMMARY:
Polymyalgia rheumatica (PMR) is a common inflammatory condition affecting elderly people and involving the girdles. The mainstay of treatment is oral glucocorticoids (GC), with the recent BSR-BHPR guidelines suggesting an initial prednisone dose comprised between 15 and 20 mg as appropriate. However, probably because of the dramatic response of PMR to GC, randomized controlled trials of treatment are lacking. As a result, there is no evidence from controlled studies on the efficacy of different initial doses or drug tapering. Objective of the study: to test if 12.5 mg prednisone/day is an adequate starting dose in polymyalgia rheumatica (PMR) and to evaluate clinical predictors of drug response.

Methods: 60 consecutive PMR patients will be treated with a starting dose of 12,5 mg/day prednisone. Clinical, laboratory, and ultrasonographic features will be recorded as possible predictors of response to prednisone. Remission is defined as disappearance of at least 75% of the signs and symptoms of PMR and normalization of ESR and CRP within the first month, a scenario allowing steroid tapering.

ELIGIBILITY:
Inclusion Criteria:

* patients with PMR, diagnosed according to the criteria of Bird et al

Exclusion Criteria:

* patients with arthritis
* patients with giant cell arteritis
* patients with Parkinson's disease
* patients with hypothyroidism
* patients with scapulohumeral periarthritis
* patients with fibromyalgia
* patients unable to cooperate

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
clinical remission within one month from the treatment initiation | 1 month
  Remission was defined as at least a 70% global improvement of the signs and symptoms of PMR and normalization of ESR and CRP within the first month, allowing steroid tapering.

SECONDARY OUTCOMES:
to evaluate demographic features as possible predictive factors of response to 12.5 mg of prednisone | 1 month
  age, sex, body weight measured at the time of the first visit were evaluated by logistic regression with response to 12.5 mg of prednison as independent variable
to evaluate characteristics of PMR as predictive factors of response to 12.5 mg of prednisone | 1 month
  duration of disease, presence of fatigue, fever, and weight loss, duration of morning stiffness were assessed in multivariate analysis with response to 12.5 mg of prednisone as independent variable
to evaluate findings at clinical examination as predictive factors of response to 12.5 mg of prednisone | 1 month
  presence of girdle tenderness, carpal tunnel syndrome, RS3PE, peripheral arthritis or tenosynovitis were studied by multivariate analysis with response to 12.5 mg prednisone as independent variable
to evaluate laboratory parameters as predictive factors of response to 12.5 mg of prednisone | 1 month
  erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), and IgM rheumatoid factor (RF) were studied by multivariate analysis with response to 12.5 mg prednisone as independent variable
to evaluate results of US as possible predictors of response to 12.5 mg prednisone | 1 month
  results of ultrasonography (US) of the shoulders were studied by multivariate analysis with response to 12.5 mh prednisone as independent variable

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Reumatologica, Dipartimento di medicina Interna, Università di Genova, Genova, Italy

REFERENCES:
- [Background] Dasgupta B, Borg FA, Hassan N, Barraclough K, Bourke B, Fulcher J, Hollywood J, Hutchings A, Kyle V, Nott J, Power M, Samanta A; BSR and BHPR Standards, Guidelines and Audit Working Group. BSR and BHPR guidelines for the management of polymyalgia rheumatica. Rheumatology (Oxford). 2010 Jan;49(1):186-90. doi: 10.1093/rheumatology/kep303a. Epub 2009 Nov 12. No abstract available. PMID 19910443
- [Derived] Cimmino MA, Parodi M, Montecucco C, Caporali R. The correct prednisone starting dose in polymyalgia rheumatica is related to body weight but not to disease severity. BMC Musculoskelet Disord. 2011 May 14;12(1):94. doi: 10.1186/1471-2474-12-94. PMID 21569559